CLINICAL TRIAL: NCT07394725
Title: Unlocking New Avenues: Azithromycin Vs Erythromycin in Pre-term, Pre-mature Rupture of Membrane Management
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: District Headquarters Teaching Hospital Sahiwal (Other)
Responsible Party: Principal Investigator, Mahpara Shaukat, Associate Professor, District Headquarters Teaching Hospital Sahiwal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130/IRV/SLMC/SWL
Record Dates: First submitted 2025-11-14; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pre-term Premature Rupture of Membranes
Keywords: Azithromycin; Erythromycin
MeSH Terms: interventions — Erythromycin; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin Group (Experimental): Participants will receive oral azithromycin as per protocol.
  Interventions: Drug: Azithromycin
- Erythromycin Group (Experimental): Participants will receive oral erythromycin as per protocol.
  Interventions: Drug: Erythromycin

INTERVENTIONS:
Drug: Erythromycin — Erythromycin 250 mg orally every 6 hours for 7 consecutive days.
  Arms: Erythromycin Group
Drug: Azithromycin — Azithromycin 500 mg orally once daily for 7 consecutive days
  Arms: Azithromycin Group

SUMMARY:
This randomized controlled trial at Sahiwal Teaching Hospital (April 2024-March 2025) compared azithromycin and erythromycin for managing preterm premature rupture of membranes (PPROM) in 250 women (28-33+6 weeks gestation). Participants received either azithromycin 500 mg once daily or erythromycin 250 mg every six hours for seven days.

DETAILED DESCRIPTION:
Background: Preterm premature rupture of membranes (PPROM) is a significant contributor to preterm births and neonatal morbidity worldwide. While erythromycin has traditionally been used for this purpose, limitations related to tolerability and dosing frequency have prompted the evaluation of alternative agents such as azithromycin.

Objective: To compare the clinical efficacy of azithromycin versus erythromycin in the management of PPROM, focusing on latency period, maternal infection rates, neonatal outcomes, and overall drug tolerability.

Methodology: This randomized controlled trial was conducted at Sahiwal Teaching Hospital from 01-04-2024 to 31-03-2025. A total of 250 pregnant women with confirmed PPROM between 28+0 and 33+6 weeks of gestation were randomly allocated into two groups: Group A oral dose of azithromycin 500mg once daily for seven days, while Group B received erythromycin 250 mg orally every six hours for seven days. Primary outcomes included latency period, incidence of chorioamnionitis, mode of delivery, and key neonatal indicators such as APGAR scores, NICU admission rates, respiratory distress syndrome (RDS), and neonatal mortality.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Aged 18 to 40 years
* Singleton pregnancy with PPROM and
* 28 weeks 0 days to 33 weeks 6 days of gestation.

Exclusion Criteria:

* Pregnancy was before 28 weeks
* Possible fetal defects
* Signs of active labor
* Major vaginal bleeding
* Signs of chorioamnionitis on arrival
* Placenta previa or placental abruption
* Allergic to macrolide antibiotics or received antibiotic treatment less than five days earlier were all excluded.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 250 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Maternal Outcome | 07 Days
  Primary Outcome Measure 1
  Name: Incidence of Clinical Chorioamnionitis
  Description:
  Clinical chorioamnionitis will be diagnosed based on predefined clinical criteria including maternal fever (≥38°C), maternal tachycardia, uterine tenderness, and foul-smelling amniotic fluid, supported by laboratory evidence of infection.
  Measurement Tool:
  Daily standardized clinical assessment and laboratory evaluation.
  Time Frame:
  Within 7 days of enrollment or until delivery, whichever occurs earlier.
  Unit of Measure:
  Number of participants diagnosed with clinical chorioamnionitis.
  Primary Outcome Measure 2
  Name: Maternal Laboratory Evidence of Infection
  Description:
  Maternal inflammatory response will be assessed using total leukocyte count (TLC) and C-reactive protein (CRP) levels to support the diagnosis of infection.
  Measurement Tool:
  Venous blood sampling for TLC and CRP.
  Time Frame:
  Measured on alternate days until delivery
Neonatal Outcomes | 07 days
  Primary Outcome Measure 3
  Name: Neonatal Birth Weight
  Description:
  Neonatal birth weight measured immediately after delivery.
  Measurement Tool:
  Calibrated digital weighing scale.
  Time Frame:
  At birth.
  Unit of Measure:
  Grams.
  Primary Outcome Measure 4
  Name: APGAR Score at 1 Minute
  Description:
  Assessment of neonatal APGAR score at 1 minute after birth.
  Measurement Tool:
  Standard APGAR scoring system.
  Time Frame:
  1 minute after birth.
  Unit of Measure:
  Score (0-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Sahiwal Teaching Hospital , Sahiwal, Sāhīwāl, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be shared due to institutional policies and concerns regarding participant confidentiality.